CLINICAL TRIAL: NCT05536362
Title: Consequences of Co-Administration of Propofol With Clonidine and Ketamine Throughout Colon Cancer Surgery
Brief Title: Propofol With Clonidine and Ketamine Throughout Colon Cancer Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nirvana Ahmed
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Colon Cancer; Post Operative Pain
MeSH Terms: conditions — Colonic Neoplasms; Pain, Postoperative | interventions — Ketamine; Clonidine

STUDY DESIGN:
Intervention Model Description: preserving hemodynamic stability, dropping post-operative pain, and dipping morphine intake
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCI propofol mixed with clonidine and ketamine (Experimental): Patient group,in which they got intravenous anaesthesia with TCI propofol mixed with clonidine and ketamine
  Interventions: Drug: TCI Propofol Injection
- TCI propofol mixed with a placebo (Experimental): Control group,in which they received intravenous anaesthesia with TCI propofol mixed with a placebo (NaCl 0.9%)
  Interventions: Drug: TCI Propofol Injection

INTERVENTIONS:
Drug: TCI Propofol Injection — To decrease postoperative pain after cancer colon surgery
  Other Names: Ketamine and clonidine

SUMMARY:
The Study Showed that combining clonidine and ketamine together can increase the likelihood of achieving a sufficient level of anaesthesia while minimizing post-operative discomfort and inflammation.

DETAILED DESCRIPTION:
This study aimd to determine whether propofol infusion combined with clonidine and ketamine is more efficient in lowering the level of IL-8, preserving operation stability, and dropping post-operative pain and morphine intake.

When paralleled to propofol alone, TIVA employing propofol infusion along with pre-operation clonidine and ketamine is effective at preserving hemodynamic stability, dropping post-operative pain, and dipping morphine intake.

For this study, sixty contestants with ASA physical status I and II, ranging in age from 35 to 65, were scheduled for colon cancer operation lasting longer than 120 minutes. This study excluded participants with a history of heart, renal and liver cell failure, allergic reaction to studied drugs, and history of epilepsy, hemodynamic instability, chronic pain, or mental illness. Using a computer-generated randomization list, the patients were randomly allocated into two groups (30 patients each).

The treated group(Group T),which got intravenous anaesthesia with TCI propofol mixed with clonidine and ketamine, the control group(Group C),which received intravenous anaesthesia with TCI propofol mixed with a placebo (NaCl 0.9%) .A third party was included in this study so neither the researchers nor the research subjects are aware of the intervention which the patients got.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I and II
2. Patients with cancer colon

Exclusion Criteria:

1. participants with a history of heart, renal and liver cell failure.
2. allergic reaction to studied drugs, and history of epilepsy,
3. hydrodynamic instability,
4. chronic pain.
5. mental illness.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Measurement of Post-operative Pain | 24-hour analgesic after surgery
  Assessment of the pain post-operatively in Pediatric patients with pain score as : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain, measured in millimetres from the left end bar to the mark placed by the kid on the 10 cm line anchored by happy faces (no pain) to sad faces (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana Elshalakany, Professor, Principal Investigator — Department of Anesthesia and I.C.U. faculty of Medicine October six university, Egypt
Locations (1):
- October 6 University Hospital, Giza, Cairo Governorate, Egypt